CLINICAL TRIAL: NCT06422351
Title: A Phase 2 Clinical Trial to Evaluate the Efficacy of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the Codon Optimized Red Cell Pyruvate Kinase (coRPK) Gene in Subjects With Pyruvate Kinase Deficiency
Brief Title: Clinical Trial to Evaluate the Efficacy of Gene Therapy for Pyruvate Kinase Deficiency
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L301-0124
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pyruvate Kinase Deficiency
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells | interventions — Methods; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Experimental): RP-L301 is a gene therapy product containing autologous genetically modified CD34+ hematopoietic stem cells containing the corrected PKLR (Pyruvate Kinase L/R) gene
  Interventions: Biological: RP-L301

INTERVENTIONS:
Biological: RP-L301 — Autologous genetically modified CD34+ hematopoietic stem cells containing the corrected PKLR (Pyruvate Kinase L/R) gene
  Other Names: Intervention/Treatment

SUMMARY:
This is an open-label Phase II trial to evaluate the efficacy of a hematopoietic cell-based gene therapy for patients with Pyruvate Kinase Deficiency (PKD).

DETAILED DESCRIPTION:
Autologous hematopoietic stem cells from mobilized peripheral blood will be transduced ex vivo (outside the body) with a lentiviral vector carrying a correct copy of the deficient PKLR (Pyruvate Kinase L/R) gene. The corrected stem cells will be infused intravenously back into the patient to correct the hematological manifestations of the disease.

ELIGIBILITY:
Inclusion Criteria

1. Pyruvate Kinase Deficiency (PKD) diagnosis with a confirmed PK-LR mutation
2. Significant anemia defined as:

   * Hemoglobin (Hb) levels <9.5 g/dL documented during 2 or more assessments in the 12 months prior to screening and either:

     1. at least 6 Red Blood Cell (RBC) transfusion episodes over the 12- month period prior to screening or
     2. at least 3 Red Blood Cell (RBC) transfusion episodes each year for 2 years prior to screening; or
   * Hemoglobin (Hb) levels <8.5 g/dL irrespective of transfusions (documented during 2 or more assessments during the prior 2 years); or
   * Hemoglobin (Hb) levels <10.0 g/dL irrespective of transfusions (documented during 2 or more assessments during the prior 2 years) and the presence of either:

     * Fatigue or energy-related symptoms limiting activities of daily living (The National Cancer Institute Common Terminology Criteria for Adverse Events v 5.0 (NCI CTCAE v5.0 grade 3)); or
     * Fatigue or energy-related symptoms limiting activities of daily living (The National Cancer Institute Common Terminology Criteria for Adverse Events v 5.0 (NCI CTCAE v5.0 grade 2)) not responsive to available medical therapy; or
     * Icterus limiting social interactions, education or work activities and not responsive to available medical therapy;
3. Subject age: age ≥8 years and ≤55 years
4. Prior splenectomy
5. Adequate cardiac, pulmonary, renal and hepatic function, as detailed in relevant exclusion criteria
6. Availability of detailed medical records, including accurate transfusion history and blood count assessments, for the prior 2 years
7. Willing and able to read and correctly understand the patient information sheet and provide consent (or informed assent for minors) regarding study participation, willing and able to comply with all study-related procedures including follow-up visits.
8. Negative serum pregnancy test for female subjects of childbearing potential.

Exclusion Criteria

1. Presence of other known causes of hemolysis (in addition to Pyruvate Kinase Deficiency (PKD)). Patients with concurrent G6PD deficiency diagnosed during pre-study evaluation may be considered for eligibility if in the opinion of the Investigator, the hemolytic anemia is the result of PKD and the Glucose-6-phosphate dehydrogenase (G6PD) deficiency is considered an incidental finding.
2. A venous thromboembolic event (VTE; i.e., pulmonary embolism or deep vein thrombosis) or arteriothromboembolic event (ATE; including unstable angina, myocardial infarction, stroke or transient ischemic attack) during the prior 12 months.
3. Evidence of bridging fibrosis, cirrhosis or active hepatitis on liver biopsy.

   1. Liver biopsy is required when liver iron concentration (LIC) is ≥15 mg/g on T2* magnetic resonance imaging (MRI) of liver.
   2. If a liver biopsy has been performed less than 6 months prior to enrollment, it does not need to be repeated.
4. Cardiac T2* <10 ms by magnetic resonance imaging (MRI) or left ventricular ejection fraction (LVEF) <45% by echocardiogram or multiple gated acquisition scan (MUGA).
5. Any evidence of severe iron overload beyond parameters stipulated in exclusion criteria 3 and 4 that, per Investigator discretion, warrants exclusion.
6. Significant medical conditions including documented HIV (human immunodeficiency virus) infection, active viral hepatitis, poorly controlled hypertension, pulmonary hypertension, cardiac arrhythmia or congestive heart failure; or arteriothromboembolic events (ATEs) (including stroke or myocardial infarction) within the 12 prior months.
7. Active hematologic or solid organ malignancy, not including non-melanoma skin cancer or another carcinoma in situ. Patients with previously resected solid organ malignancies or definitively treated hematologic malignancies may be eligible if there has been no evidence of active malignancy during the prior 3 years.
8. Uncontrolled seizure disorder.
9. Hepatic dysfunction as defined by Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5× the upper limit normal (ULN).
10. Renal dysfunction defined as serum creatinine >upper limit normal (ULN). Patients with creatinine above ULN may be eligible pending documentation of a glomerular filtration rate ≥60 mL/min/1.73m2 as calculated by Modification of Diet in Renal Disease equation (Stevens 2006), or 24-hour urine collection.
11. Pulmonary dysfunction as defined by either:

    1. Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection) OR
    2. Clinically significant pulmonary disease that may impair ability to tolerate study procedures and treatments.
12. Any medical or other contraindication for leukapheresis as determined by the treating Investigator.
13. Any medical or psychiatric condition that in the opinion of the Investigator renders the patient unfit for trial participation or at higher than acceptable risk for participation.
14. Poor functional status evidenced by Karnofsky Index <70 in subjects ≥16 years old and Lansky Play-Performance Scale <70 in subjects <16 years old.
15. Participation in another clinical trial with an investigational drug within 14 days before the informed consent signature. Participation in observational studies is allowed. Patients who are receiving mitapivat in non-investigational settings are eligible provided they discontinue mitapivat at least 90 days prior to the start of mobilization.
16. Pregnant women or women with a positive serum pregnancy test at screening or breast feeding or planning to become pregnant within the next 24 months. Female participants or female partners of male participants not willing to use highly effective contraceptive methods during the complete study period.
17. Previous allogeneic or other hematopoietic stem cell transplant.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Anemia | 12 months post-infusion
  Hemoglobin (Hb) level increase of ≥1.5g/dL at 12 months post-infusion, compared to baseline.

SECONDARY OUTCOMES:
Durability Improvement anemia sustained | 24 months post-infusion
  Time to Hemoglobin level increase of ≥1.5g/dL post-infusion, compared to baseline.
Resolution of anemia | 12 months post-infusion
  Hemoglobin level within normal range (≥ lower limit of normal) at 12 months post-infusion.
Reduction of transfusion requirements | 12 months post-infusion
  * a: ≥50% reduction in Pyruvate Kinase Deficiency (PKD)-related Red Blood Cells (RBC) transfusion requirements in the 12 months post-infusion, relative to the annualized event rate for 24 months prior to enrollment; or,
  * b: Absence of PKD-related RBC transfusion requirements in the 12 months post-infusion.
Improvements of hemolysis parameters (bilirubin) | 12 months post-infusion
  Improvements in bilirubin, each evaluated at 12 months post-infusion, compared to baseline.
Improvements of hemolysis parameters (Lactate Dehydrogenase (LDH)) | 12 months post-infusion
  Improvements in Lactate Dehydrogenase (LDH), each evaluated at 12 months post-infusion, compared to baseline.
Improvements of hemolysis parameters (erythropoietin) | 12 months post-infusion
  Improvements in erythropoietin, each evaluated at 12 months post-infusion, compared to baseline.
Improvements of hemolysis parameters (reticulocyte) | 12 months post-infusion
  Improvements in reticulocyte, each evaluated at 12 months post-infusion, compared to baseline.
Peripheral blood genetic correction | 12 months post-infusion
  Genetic correction demonstrated by vector copy number (VCN) of 0.1 in Peripheral Blood mononuclear cells, evaluated at 12 months post-infusion.
Improvement in fatigue | 12 months post-infusion
  Improvement in fatigue as compared with baseline, as assessed by:
  * Age ≥18: FACIT Fatigue; or,
  * Age <18: PROMIS Fatigue Short Form 10a
Improvement in dyspnea | 12 months post-infusion
  Improvement in Pyruvate Kinase Deficiency symptoms, compared with baseline, as assessed by:
  * PROMIS Dyspnea Severity SF10; or,
  * Dyspnea severity
Improvement in jaundice | 12 months post-infusion
  Improvement in Pyruvate Kinase Deficiency symptoms, compared with baseline, as assessed by:
  * jaundice severity evaluated at 12 months post-infusion; or,
  * and jaundice severity
Safety and tolerability of RP-L301 | 24 months post-infusion
  Incidence, type, severity, frequency, time to onset, and duration of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), clinical laboratory abnormalities, and adverse events of special interest (AESIs).
Evaluate durable resolution of anemia | 24 months post-infusion
  Hemoglobin (Hb) level within normal range (≥ lower limit of normal).
Evaluate durable resolution of transfusion requirements (where relevant). | 24 months post-infusion
  1. ≥50% reduction in Pyruvate Kinase Deficiency (PKD)-related Red Blood Cell (RBC) transfusion requirements in the 24 months post-infusion, relative to the annualized event rate for 24 months prior to enrollment; or,
  2. Absence of PKD-related RBC transfusion requirements in the 24 months post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ami Shah, MD, Principal Investigator — Stanford University; Julian Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús; José Luis López Lorenzo, MD, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz; Elieen Nicoletti, MD, Study Director — Rocket Pharmaceuticals Inc.
Locations (3):
- Stanford University, Palo Alto, California, United States
- Spain (2):
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No